CLINICAL TRIAL: NCT02841956
Title: Reducing Duration of Untreated Psychosis Through Rapid Identification and Engagement
Acronym: DUP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 608950; R01MH104235 (NIH)
Record Dates: First submitted 2016-06-29; First posted 2016-07-22 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders | interventions — Educational Status; Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Electronic Screen + Education (Phase 1) (Experimental): Electronic screening of participants and targeted education of providers according to standard EDAPT model.
  Interventions: Other: Electronic Screen + Education (Phase 1)
- Targeted Provider Education (Phase 1) (Active Comparator): Targeted education of providers according to standard EDAPT model.
  Interventions: Other: Targeted Provider Education (Phase 1)
- Community Mobile Engagement (Phase 2) (Experimental): Clinical intake interviews take place via videoconference at a location in the community convenient for the participant.
  Interventions: Other: Community Mobile Engagement (Phase 2)
- Clinic based Engagement (Phase 2) (Active Comparator): Clinical intake interviews take place at the EDAPT clinic.
  Interventions: Other: Clinic based Engagement (Phase 2)

INTERVENTIONS:
Other: Electronic Screen + Education (Phase 1) — PHASE 1 Electronic Screening Arm + Targeted Education: Referral sources will receive the same standard targeted education as active comparator. In addition, the PQ-B (a 21 item screening questionnaire) will be administered to all patients at their first visit to the referral sites (e.g. intake) via an android tablet provided to the site for ease of administration and scoring. The investigators will provide multiple tablets per site so that the screening is available for more than one individual simultaneously and can be completed in any appropriate location. The investigators will allow paper-and-pencil administration for situations where it is more appropriate (e.g. emergency room).
  Arms: Electronic Screen + Education (Phase 1)
Other: Targeted Provider Education (Phase 1) — PHASE 1 Targeted Education Intervention: EDAPT standard targeted provider education1 focuses on increasing awareness about the signs of early psychosis & building collaborative relationships with community members so community members see EDAPT as a rapid, effective source of help. It consists of a 2-hour workshop describing: 1) how to identify specific early symptoms & changes associated with the onset of psychotic illness, 2) the benefits of early intervention on treatment outcomes in psychosis, 3) the structure, philosophy & treatment model of the EDAPT Clinic, and 4) procedures for expeditious referral to our program. Case-based vignettes are reviewed to ensure understanding of the key symptoms.
  Arms: Targeted Provider Education (Phase 1)
Other: Community Mobile Engagement (Phase 2) — PHASE 2 Community-based Mobile Engagement: Clinical assessment appointments will take place at the EDAPT clinic or within the community, wherever the individual would prefer. With patients deemed eligible for EDAPT services, the EDAPT clinician will obtain vitals and contact the EDAPT psychiatrist with a telemedicine-enabled laptop to complete the psychiatric evaluation remotely. The psychiatrist will prescribe medications and order labs, as indicated. The EDAPT clinician will follow up with the individual within 5 days to determine if the prescribed medication regimen has started.
  Arms: Community Mobile Engagement (Phase 2)
Other: Clinic based Engagement (Phase 2) — PHASE 2 Clinic-based Engagement: The clinical assessment appointment will be completed within the EDAPT clinic. If deemed eligible for EDAPT services, the individual will be scheduled for a clinic-based appointment with the EDAPT psychiatrist within 5 days, who will prescribe medications and order labs as indicated. The EDAPT clinician will follow up with the individual within 5 days of the psychiatric evaluation (by phone or in the clinic) to determine if the prescribed medication regimen has started.
  Arms: Clinic based Engagement (Phase 2)

SUMMARY:
Reducing Duration of Untreated Psychosis (DUP) is a primary goal for improving long-term outcomes in young people with a first episode of psychosis (FEP). The "standard of FEP care" within the US focuses on targeted provider education regarding signs and symptoms of early psychosis to motivate patient referrals to FEP services, followed by initiation of services within largely clinic-based settings Experience at the Early Diagnosis and Preventive Treatment (EDAPT) FEP specialty program at U.C. Davis in Sacramento has identified two important bottlenecks to reducing DUP, consistent with reports in the literature from other FEP clinics. These are 1) delays in the identification of psychotic symptoms by referral sources, and 2) delays or disruptions of patient engagement in specialty FEP care. Building upon a comprehensive and established referral network of 20 sites across the Sacramento area (schools/universities, ER/inpatient hospitals, outpatient mental health, primary care), the investigators will address delays in patient identification and engagement using a two-phase, cluster randomized design. The investigators will consecutively test the impact of two interventions to reduce DUP, defined in this RFA as time from first onset of psychotic symptoms to engagement in FEP specialty care. To address identification delays, the investigators will examine the use of standard targeted provider education plus novel technology-enhanced screening compared to standard targeted provider education alone, testing the hypothesis that the education plus technology-enhanced screening will identify more patients, earlier in their illness. To address engagement delays, the investigators will compare the use of a mobile community-based, telepsychiatry-enhanced engagement team to standard clinic-based procedures for intake, engagement and initiation of treatment, to test the hypothesis that the mobile approach facilitates earlier and more stable engagement, thereby reducing DUP. The proposed work will provide new specific evidence-based practices for reducing DUP and improving outcomes through specialty care of individuals with a first episode of psychosis.

ELIGIBILITY:
Inclusion criteria:

Meet DSM-IV criteria for a diagnosis of affective or nonaffective psychosis.

Exclusion criteria:

1. Duration of psychosis > 2 years
2. Current substance dependence
3. Neurological illness or injury leading to psychotic symptoms
4. Only substance induced psychotic symptoms
5. Documented IQ < 70
6. Lack of English fluency

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 427 (Actual)
Dates: Start 2014-09; Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Days of active psychosis between onset of illness and identification for care (Duration of untreated psychosis) | Day 1

SECONDARY OUTCOMES:
Rates of patient enrollment in first episode psychosis care | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis Early Diagnosis and Preventative Treatment (EDAPT) Clinic, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Niendam TA, Loewy R, Savill M, Delucchi KL, Lesh TA, Ragland JD, Bolden K, Skymba HV, Gobrial S, Meyer MS, Pierce KM, Rosenthal A, Fedechko TL, Tully LM, Tryon VL, Goldman H, Cress RD, Kravitz RL, Carter CS. Effect of Technology-Enhanced Screening in Addition to Standard Targeted Clinician Education on the Duration of Untreated Psychosis: A Cluster Randomized Clinical Trial. JAMA Psychiatry. 2023 Feb 1;80(2):119-126. doi: 10.1001/jamapsychiatry.2022.4436. PMID 36598770
- See also: UC Davis Early Psychosis Programs — http://earlypsychosis.ucdavis.edu